CLINICAL TRIAL: NCT01884155
Title: Safety and Efficacy of Allogeneic Umbilical Cord Blood Therapy for Patients With Stroke
Brief Title: Allogeneic Umbilical Cord Blood Therapy for Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MinYoung Kim, M.D. (Other)
Responsible Party: Sponsor-Investigator, MinYoung Kim, M.D., Professor, Bundang CHA Hospital
Organization: Bundang CHA Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCBStroke
Record Dates: First submitted 2013-06-19; First posted 2013-06-21 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: allogeneic cord blood for stroke patients
Oversight: Data Monitoring Committee: No

ARMS (1):
- Allogeneic umbilical cord blood therapy (Experimental): Allogeneic umbilical cord blood therapy
  Interventions: Procedure: Allogeneic umbilical cord blood therapy

INTERVENTIONS:
Procedure: Allogeneic umbilical cord blood therapy

SUMMARY:
This open label trial is conducted to investigate the efficacy and safety of allogeneic umbilical cord blood (UCB) therapy for patients with stroke.

DETAILED DESCRIPTION:
Stroke is one of the most common etiologies causing disability in developed countries. There remains no proven treatments except tissue plasminogen activator currently. Based on promising results of cell therapy in animal stroke models, efforts to apply cell therapy for patients with stroke has been made. UCB possess various stem or progenitor cells and is known to secrete neurotrophic factors to repair injured brain. This clinical research aims to determine the safety and efficacy of allogeneic UCB for stroke.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke
* Onset duration over 12 months
* Hemisphere lesions except brain stem and cerebellar lesions
* National Institute Health Stroke Scale: 10 to 15

Exclusion Criteria:

* Possibility of hypersensitivity drugs used in this study
* Uncontrolled hypertension or cardiovascualr diseases
* Malignant cancer
* Renal or hepatic dysfunction (Consultation to specialist in nephrology or gastroenterology in case of renal or hepatic dysfunction)
* Severe pulmonary dysfunction
* Traumatic brain injury
* Lack of matched UCB

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-06; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes in Balance | Baseline - 1 month - 3 months - 6 months - 12 months

SECONDARY OUTCOMES:
Changes in Mobility | Baseline - 1 month - 3 months - 6 months - 12 months
Changes in Muscle strength and Spasticity | Baseline - 1 month - 3 months - 6 months - 12 months
Changes in Activities of Daily Living | Baseline - 1 month - 3 months - 6 months - 12 months
Changes in Function of Upper extremity | Baseline - 1 month - 3 months - 6 months - 12 months
Changes in Hand function | Baseline - 1 month - 3 months - 6 months - 12 months
Changes in Visual perception | Baseline - 1 month - 3 months - 6 months - 12 months
Changes in Cognition | Baseline - 1 month - 3 months - 6 months - 12 months
Changes in Language | Baseline - 1 month - 3 months - 6 months - 12 months
Changes in Sensory function | Baseline - 1 month - 3 months - 6 months - 12 months
Changes in Brain structure | Baseline - 12 months
Changes in Brain glucose metabolism | Baseline - 12 months
Changes in Neural activity | Baseline - 6 months - 12 months
Monitoring Adverse Events | Baseline - 1 month - 3 months - 6 months - 12 months

CONTACTS AND LOCATIONS:
Overall Officials: MinYoung Kim, M.D., Ph.D., Principal Investigator — CHA University
Locations (1):
- CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do, South Korea